CLINICAL TRIAL: NCT03698240
Title: Mindfulness-based Program for Children With Disruptive Behavior Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Pisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIND-DBD
Record Dates: First submitted 2018-06-20; First posted 2018-10-05 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-01

CONDITIONS: Disruptive Behavior Disorder; Oppositional Defiant Disorder; Attention Deficit and Disruptive Behavior Disorders
Keywords: Mindfulness; ADHD; Oppositional Defiant Disorder
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based program (Experimental): Children and parents receive the program
  Interventions: Behavioral: Mindfulness-based program
- Waiting-list (No Intervention): Children and parents receive no-interventions.

INTERVENTIONS:
Behavioral: Mindfulness-based program — The program includes 9 mindfulness-based sessions for children and their parents.
  Other Names: Fiore dentro
  Arms: Mindfulness-based program

SUMMARY:
The present RCT study investigates whether combined mindfulness program for children and their parents was beneficial for Italian children, aged 8-12, with disruptive behavior diagnosis (DBD). The study tests the program effects on children's behavioral difficulties in school and home contexts; children's and parents' mindfulness abilities; children's impulsiveness; and parents' stress. The study include a sample of 50 children randomly allocate to the intervention or to the control condition (wait-list control sample). Repeated measures of children's and parents' and teachers' reported measures will be used.

ELIGIBILITY:
Inclusion Criteria:

* Disruptive Behavior primary diagnosis

Exclusion Criteria:

* IQ < 80
* ASD diagnosis
* ongoing other interventions

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in behavioral problems at school | One week before the start of the intervention, one week after the end of the intervention.
  Strengths and Difficulties Questionnaire Strength and Difficulties Questionnaire (SDQ) is one of the most frequently used behavioral rating scale in educational, research, and clinical settings for assessing emotional and behavioral patterns in childhood. This 25-item questionnaire measures psychological adjustment in 3- to 16-year-olds in five subdomains. Of these, four subscales measure difficulties (conduct problems, hyperactivity, emotional problems, and peer relational problems), while the fifth measures strengths (prosocial behavior). There are three versions of the scale (a parent, teacher, and self-report).
Change in Aggressive behaviors | One week before the start of the intervention, one week after the end of the intervention.
  Modified Overt Aggression Scale The MOAS (Kay et al., 1988) is a clinician administered scale that measures four types of overt aggression over the past week: verbal aggression, physical aggression against property, auto-aggression, and physical aggression against other people.
Change in Behavioral problems at home | One week before the start of the intervention, one week after the end of the intervention.
  Child Behavior Check List It is a 118 item standardized format, completed by parents for recording behavioural problems and skills in children 6 to 18 years of age. The 118 behaviour problem items are aggregated in eight different subscales related to both Internalizing and Externalizing domains.
Change in impulsiveness | One week before the start of the intervention, one week after the end of the intervention.
  Matching Familiar (MF-20) test from Italian Battery for ADHD (Marzocchi, Re, & Cornoldi, 2010). In the Matching Familiar Figures (MF) test, participants are shown a figure and are asked to find the matching one among six choices. This task measures the children's impulsiveness. The MF test includes 20 items. Clinicians sum children's score in accuracy and latency time to arrive at one reported value, that is the children's impulsiveness score.
Change in sustained attention capacities | One week before the start of the intervention, one week after the end of the intervention.
  Bells Test Revised The Bells Test revised (Biancardi & Stoppa, 1997) is a test for the evaluation of sustained attention in children. The test is an adaptation of Gauthiers's Bell Test used to assess neglect in adults. The Bells Test has been modified in order to make it suitable to research in developmental age. Items are organized in four different pages, which include each 35 bells. Speed and Accuracy in selecting the target stimuli (bells) are assessed. The Speed score refers to the number of bells found by the child in the first 30 seconds of the task, while the Accuracy score refers to the total number of bells found during the whole task (120 seconds).

SECONDARY OUTCOMES:
Change in children's mindfulness abilities | One week before the start of the intervention, one week after the end of the intervention.
  Child and Adolescent Mindfulness Measure The CAMM is a recently developed questionnaire that assesses present-moment awareness and non-judgmental, non-avoidant responses to thoughts and feelings in children and adolescents (i.e., "I keep myself busy so I don't notice my thoughts or feelings"), and the ten items are rated on a fivepoint scale. The CAMM has been shown to be reliable (α= 0.81), and positive correlations have been shown with quality of life, social skills, and academic performance. Negative correlations were shown with somatic complaints, internalizing, and externalizing symptoms (Greco et al. 2011).
Change in parents' mindfulness abilities | One week before the start of the intervention, one week after the end of the intervention.
  Five Facet Mindfulness Questionnaire The FFMQ is a 39-item questionnaire that measures five facets of mindfulness (Baer et al., 2006): observing (8 items, e.g., I notice the smells and aromas of things), describing (8 items, e.g., I'm good at finding the words to describe my feelings), acting with awareness (8 items; e.g., I am easily distracted), nonjudging (8 items, e.g., I criticize myself for having irrational or inappropriate emotions), and nonreactivity (7 items; e.g., I watch my feelings without getting lost in them). Participants were asked to rate the degree to which each statement is true for them. Items were scored on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Facet scores were computed by summing the scores on the individual items. Facet scores range from 8 to 40 (except for the nonreactivity facet, which ranges from 7 to 35), with higher scores indicating more mindfulness.
Change in children's anxiety traits | One week before the start of the intervention, one week after the end of the intervention.
  Multidimensional Anxiety Scale for Children The Multidimensional Anxiety Scale for Children (MASC) is a 39-item, 4-point Likert self-report scale that robustly represents the factor structure of anxiety in children aged 8 to 18 years. MASC main and subfactors include (a) physical symptoms (tense/restless and somatic/autonomic), (b) harm avoidance (anxious coping and perfectionism), (c) social anxiety (humiliation/rejection and public performance fears), and (d) separation anxiety.
Change in parenting practices | One week before the start of the intervention, one week after the end of the intervention.
  Alabama Parenting Questionnaire The APQ is a 42-item measure on which parents were asked to indicate the frequency with which they implemented a range of parenting practices on a 5-point scale, ranging from 1 (never) to 5 (always). The subfactors include: a) positive parenting, b) parental involvement, c) inconsistent discipline, d) corporal punishment.
Change in parents' stress | One week before the start of the intervention, one week after the end of the intervention.
  Parenting Stress Index The PSI-SF is a 36- item questionnaire designed to measure stress in the parent-child system and identify those families most in need of follow-up services. The PSI-SF consists of three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Each subscale consists of 12 items rated from 1 (strongly disagree) to 5 (strongly agree). Subscale scores therefore range from 12 to 60, whereas the total score ranges from 36 to 180. High scores on the subscales and PSI-SF total score indicate greater levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Muratori, Principal Investigator — IRCCS Stella Maris
Locations (1):
- IRCCS Stella Maris, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No